CLINICAL TRIAL: NCT02784483
Title: Pilot Study Of Anti-Programmed Death Ligand-1 (Anti-PD-L1, Atezolizumab) In Asymptomatic Myeloma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Based on FDA requirements
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1511016813
Record Dates: First submitted 2016-05-24; First posted 2016-05-27 (Estimated); Last update posted 2020-03-03 (Actual); Status verified 2020-02

CONDITIONS: Asymptomatic Myeloma
MeSH Terms: conditions — Smoldering Multiple Myeloma | interventions — atezolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Atezolizumab (1200mg via IV infusion) (Experimental)
  Interventions: Drug: Atezolizumab (1200mg via IV infusion)

INTERVENTIONS:
Drug: Atezolizumab (1200mg via IV infusion) — Patients will get atezolizumab every 21 days for up to 1 year

SUMMARY:
The purpose of this pilot study is to gain initial insights into the biologic and clinical effects of Atezolizumab in patients with Asymptomatic Multiple Myeloma (AMM). The data may provide novel insights into anti-PDL-1-induced immunologic changes, which could potentially be relevant to its future development in Multiple Myeloma (MM) and other indications.

ELIGIBILITY:
INCLUSION CRITERIA:

Patients must meet the following criteria for study entry:

* All patients must sign an Informed Consent Form (ICF) approved by Institutional Review Board, and express ability and willingness to comply with the requirements of the study protocol.
* Patients must meet criteria for high risk AMM defined as:

  * Bone marrow plasma cells ≥ 10% and/or levels of monoclonal protein (M-protein) >3 g/dL and
  * Abnormal FLC ratio and absence of end organ damage (CRAB) defined as: lytic bone lesions on skeletal survey, calcium ≥ 11mg/dl, hemoglobin value of >2 g/100 ml below the lower limit of normal or a hemoglobin value <10 g/100 ml and renal insufficiency(serum creatinine >0.173 mmol/l) Note: Patients with BMPC > 60%, serum free light chain ratio >100, or known to have 2 or greater focal lesions on MRI and are clinically felt to require therapy will not be included.
* Measurable disease defined by: M-spike >1 g/dL, or Bence Jones protein > 200 mg/24 hours by urine protein electrophoresis or involved serum free light chain (FLC) >10 mg /dl
* Adequate hematologic and end organ function, defined by the following laboratory results obtained within 28 days prior to the first study treatment (Cycle 1, Day 1):

  * ANC ≥ 1500 cells/ µL
  * WBC counts > 2500/ µL
  * Lymphocyte count ≥ 300/ µL
  * Platelet count ≥ 75,000/ µL
  * Total bilirubin within normal range
  * AST and ALT within normal range
  * Serum creatinine within normal range or creatinine clearance ≥ 60 mL/min on the basis of the Cockcroft-Gault glomerular filtration rate estimation:

    (140 - age) x (weight in kg) x (0.85 if female) / 72 x (serum creatinine in mg/dL)
* For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods that result in a failure rate of < 1% per year during the treatment period and for at least 90 days after the last dose of study drug.

  * A woman is considered to be of childbearing potential if she is postmenarcheal, has not reached a postmenopausal state (≥ 12 continuous months of amenorrhea with no identified cause other than menopause), and has not undergone surgical sterilization (removal of ovaries and/or uterus).
  * Examples of contraceptive methods with a failure rate of < 1% per year include bilateral tubal ligation, male sterilization, established, proper use of hormonal contraceptives that inhibit ovulation, hormone-releasing intrauterine devices, and copper intrauterine devices.
  * The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not acceptable methods of contraception.
* For men: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures and agreement to refrain from donating sperm, as defined below:

  * With female partners of childbearing potential or pregnant female partners, men must remain abstinent or use a condom during the treatment period and for at least 90 days after the last dose of study drug. Men must refrain from donating sperm during this same period.
  * The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not acceptable methods of contraception.

EXCLUSION CRITERIA:

Patients who meet any of the following criteria will be excluded from study entry.

General Exclusion Criteria:

* Any approved anticancer therapy, including chemotherapy, hormonal therapy, or radiotherapy, within 3 weeks prior to initiation of study treatment; however, the following are allowed:

  * Herbal therapy > 1 week prior to Cycle 1, Day 1 (herbal therapy intended as anticancer therapy must be discontinued at least 1 week prior to Cycle 1, Day 1)
* AEs from prior anticancer therapy that have not resolved to Grade ≤ 1 except for alopecia
* Known liver disease, including active viral, alcoholic, or other hepatitis; cirrhosis; fatty liver; and inherited liver disease
* Known hypersensitivity to Chinese hamster ovary cell products or other recombinant human antibodies
* Inability to comply with study and follow-up procedures
* History of active autoimmune disease, including but not limited to systemic lupus erythematosus, rheumatoid arthritis, type 1 diabetes mellitus, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjögren's syndrome, Bell's palsy, Guillain-Barré syndrome, multiple sclerosis, autoimmune thyroid disease, vasculitis, glomerulonephritis or autoimmune related dermatologic disease
* History of idiopathic pulmonary fibrosis, pneumonitis (including drug induced), organizing pneumonia (i.e., bronchiolitis obliterans, cryptogenic organizing pneumonia, etc.).
* Any other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or render the patient at high risk from treatment complications
* History of HIV infection or known active hepatitis B (chronic or acute) or hepatitis C infection

  * Patients with past or resolved hepatitis B infection (defined as having a negative hepatitis B surface antigen [HBsAg] test and a positive anti-HBc [antibody to hepatitis B core antigen] antibody test) are eligible.
  * Patients positive for hepatitis C virus (HCV) antibody are eligible only if polymerase chain reaction (PCR) is negative for HCV RNA.
* Active tuberculosis requiring therapy.
* Severe infections within 4 weeks prior to Cycle 1, Day 1, including but not limited to hospitalization for complications of infection, bacteremia, or severe pneumonia
* Major surgical procedure within 28 days prior to Cycle 1, Day 1 or anticipation of need for a major surgical procedure during the course of the study
* Administration of a live, attenuated vaccine within 4 weeks before Cycle 1, Day 1 or anticipation that such a live, attenuated vaccine will be required during the study

  * Influenza vaccination should be given during influenza season only. Patients must not receive live, attenuated influenza vaccine (e.g., FluMist™) within 4 weeks prior to Cycle 1, Day 1 or at any time during the study.
* Malignancies other than myeloma within 5 years prior to Cycle 1, Day 1, with the exception of those with a negligible risk of metastasis or death and with expected curative outcome (such as adequately treated carcinoma in situ of the cervix, basal or squamous cell skin cancer, localized prostate cancer treated surgically with curative intent, or ductal carcinoma in situ treated surgically with curative intent) or undergoing active surveillance per standard-of-care management (e.g., chronic lymphocytic leukemia Rai Stage 0, prostate cancer with Gleason score ≤ 6, and prostate-specific antigen [PSA] ≤ 10 mg/mL, etc.).

Medication-Related Exclusion Criteria:

* Prior treatment with anti-PD-1, or anti-PD-L1 therapeutic antibody or pathway targeting agents.
* Treatment with another investigational agent within 4 weeks prior to Cycle 1, Day 1 (or within five half lives of the investigational product, whichever is longer)
* Treatment with systemic immunosuppressive medications (including but not limited to prednisone, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor [anti-TNF] agents) within 2 weeks prior to Cycle 1, Day 1.

  * Patients who have received acute, low dose, systemic immunosuppressant medications (e.g., a one-time dose of dexamethasone for nausea) may be enrolled.
  * The use of inhaled corticosteroids and mineralocorticoids (e.g., fludrocortisone) for patients with orthostatic hypotension or adrenocortical insufficiency is allowed.
* History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2017-02-10 (Actual); Primary Completion 2017-09-15 (Actual); Study Completion 2019-04-22 (Actual)

PRIMARY OUTCOMES:
Prevalence of anti-SOX2 reactive T cells after Anti-PDL1 therapy | Up to 1 year
  Presence or absence of SOX2 cells before and after anti-PDL1 therapy followed up to 1 year will be measured using antigen dependant stimulation.

CONTACTS AND LOCATIONS:
Overall Officials: Noffar Bar, MD, Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bar N, Costa F, Das R, Duffy A, Samur M, McCachren S, Gettinger SN, Neparidze N, Parker TL, Bailur JK, Pendleton K, Bajpai R, Zhang L, Xu ML, Anderson T, Giuliani N, Nooka A, Cho HJ, Raval A, Shanmugam M, Dhodapkar KM, Dhodapkar MV. Differential effects of PD-L1 versus PD-1 blockade on myeloid inflammation in human cancer. JCI Insight. 2020 Jun 18;5(12):e129353. doi: 10.1172/jci.insight.129353. PMID 32427579